CLINICAL TRIAL: NCT02193633
Title: TAX-TORC: a Phase I Multi-centre Trial of the Combination of AZD2014 (dual MTORC1 and MTORC2 Inhibitor) and Weekly Paclitaxel in Patients with Solid Tumours.
Brief Title: A Phase I Trial of the Combination of AZD2014 and Weekly Paclitaxel.
Acronym: TAX-TORC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Institute of Cancer Research, United Kingdom (Other); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCR3667; 2012-003896-20 (EudraCT Number)
Record Dates: First submitted 2013-06-10; First posted 2014-07-17 (Estimated); Last update posted 2024-09-26 (Actual); Status verified 2020-02

CONDITIONS: Advanced Cancer
MeSH Terms: interventions — vistusertib; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AZD2014 3 on/4 off & weekly paclitaxel (Experimental): 3 days on, 4 days off AZD2014 BD administered orally Days 1-3 each week in combination with paclitaxel administered via IV infusion on Day 1 each week, in 7-week cycles (6 weeks treatment followed by 1 week rest).
  Interventions: Drug: AZD2014 3 on/4 off & weekly paclitaxel
- AZD2014 2 on/5 off & weekly paclitaxel (Experimental): AZD2014 BD administered orally Days 1-2 each week in combination with paclitaxel administered via IV infusion on Day 1 each week, in 7-week cycles (6 weeks treatment followed by 1 week rest).
  Interventions: Drug: AZD2014 2 on/5 off & weekly paclitaxel

INTERVENTIONS:
Drug: AZD2014 3 on/4 off & weekly paclitaxel — AZD2014 3 days on, 4 days off + weekly paclitaxel
  Other Names: AZD2014; AZD2014 3 days on, 4 days off; Paclitaxel
  Arms: AZD2014 3 on/4 off & weekly paclitaxel
Drug: AZD2014 2 on/5 off & weekly paclitaxel — AZD2014 2 days on, 5 Days off + weekly paclitaxel
  Other Names: AZD2014; AZD2014 2 days of, 5 days off; Paclitaxel
  Arms: AZD2014 2 on/5 off & weekly paclitaxel

SUMMARY:
This is a Phase I study to evaluate the safety and toxicity profile of AZD2014, a novel anticancer agent, in combination with paclitaxel.

AZD2014 will be given orally, twice daily at a starting dose of 25 mg per day for 3 days on, 4 days off with a weekly infusion of 80 mg of paclitaxel for 6 weeks followed by a treatment break of one week, therefore each cycle will be 7 weeks long. Cohorts of three patients will be treated at this dose of AZD2014 and then at 50mg and 75 mg providing is it safe to do so. Once we have determined the maximum tolerated dose (MTD) using the 3 days on, 4 days off schedule of AZD2014, patients will be given AZD2014 2 days on, 5 days with their paclitaxel infusion. Patients will be enrolled in cohorts of three to evaluate three escalating doses of AZD2014 to determine the MTD for the 2 days on, 5 days off schedule.

On completion of the dose escalation phase of the study patients with ovarian cancer and squamous cell lung cancer will be treated at the MTD established for each dosing schedule. A minimum of 10 ovarian cancer patients and 15 squamous cell lung patients will be enrolled to the 3 days on, 4 days off schedule. Whilst a minimum of 10 squamous cell cancer patients will be enrolled to the 2 days on, 5 days off schedule to further assess the tolerability of the combination of AZD2014 and paclitaxel.

DETAILED DESCRIPTION:
This is a multi-centre, Phase I clinical trial of the combination of AZD2014 and weekly paclitaxel.

Two intermittent BD dosing schedules of AZD2014 in combination with paclitaxel will be evaluated. The 3 days on 4 days off schedule will examine 3 continuous days of AZD2014 per week in combination with weekly paclitaxel. The 2 days on 5 days off schedule will examine 2 sequential days of AZD2014 dosing in combination with weekly paclitaxel. For both schedules, a dose escalation 3+3 design will be used to establish the MTD and the recommended Phase II dose. Approximately 15 patients with solid tumours will be entered into each schedule during the dose escalation of this phase.

The expansion part of the trial will be used to further assess the tolerability of AZD2014 in combination with weekly paclitaxel. For the 3 days on 4 days off schedule 10 patients with ovarian cancer and 15 patients with squamous lung cancer will be enrolled and treated at the MTD established from the dose escalation phase. Accrual to these expansion arms may commence as soon as the MTD is determined and proceed in parallel with the dose escalation phase of the 2 days on 5 days off schedule. Once the MTD has been determined for the 2 days on 5 days off schedule 15 patients with squamous lung cancer may be enrolled.

Determination of the MTD and decision to enter the expansion phase for each schedule will be made by the Safety Review Committee (SRC) taking into consideration the safety data and available PK/PD data.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically proven solid tumour.refractory to conventional treatment, or for which no conventional therapy exists or is declined by the patient, or where treatment with paclitaxel is an appropriate treatment option. Patients enrolled in the expansion phase must have recurrent ovarian, fallopian tube or primary peritoneal cancer only.
2. Patients who have had conventional treatment and where paclitaxel is appropriate. In instances where paclitaxel is appropriate but the patients has not already received it the patient may be enrolled after discussion between the referring oncologist and Principal Investigator.
3. Life expectancy of at least 12 weeks
4. ECOG performance status of 0-1
5. Females should be using adequate contraceptive measures, should not be breast feeding and must have a negative pregnancy test prior to start of dosing if of child-bearing potential or must have evidence of non-child-bearing potential
6. Male patients should be willing to use barrier contraception i.e., condoms
7. Measurable or evaluable disease. Patients enrolled in the expansion phase should have measurable disease by RECIST v1.1 criteria
8. Haematological and biochemical indices within the ranges shown below. These measurements must be performed within one week (Day -7 to Day 1) before the patient goes in the trial.

   * Haemoglobin (Hb)≥ 9.0 g/dL
   * Absolute neutrophil count ≥ 1.5 x 109/L
   * Platelet count ≥ 100 x 109/L
   * Serum bilirubin ≤ 1.5 x upper limit of normal (ULN)
   * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST)≤ 2.5 x (ULN) if no demonstrable liver metastases or ≤ 5 times ULN in the presence of liver metastases
   * Alkaline phosphatase (ALP)< 5 x ULN
   * Creatinine Clearance ≥ 50 mL/min (uncorrected value)OR Serum creatinine ≤ 1.5 x ULN
   * Fasting glucose ≤ 125 mg/dL (7 mmol/L)
   * Erythrocyte-HbA1c ≤ 59 mmol/mol
9. 18 years or over
10. Written (signed and dated) informed consent and be capable of co-operating with treatment and follow-up

Exclusion Criteria:

1. Radiotherapy (except for palliative reasons), chemotherapy, endocrine therapy, or immunotherapy during the previous 3 weeks (4 weeks for investigational medicinal products and 6 weeks for nitrosoureas and Mitomycin-C) before treatment.

   N.B. Exceptions to this are patients receiving weekly taxol as standard of care who have not had a partial or complete response after 6 to 12 weekly doses. Those patients should discontinue their weekly taxol treatment and may be enrolled to the dose expansion phase without a wash out period.
2. CTCAE Grade 1 or higher toxicities from previous systemic anticancer therapy prior to the first dose of study treatment (with the exception of alopecia)
3. Known leptomeningeal involvement, brain metastases or spinal cord compression
4. Known hypersensitivity (>Grade 2) to taxanes, drugs containing Cremophor, AZD2014 or structurally/chemically similar drugs
5. Unresolved bowel obstruction
6. Current refractory nausea and vomiting, chronic gastrointestinal disease, inability to swallow formulated product or previous significant bowel resection that would preclude adequate absorption of AZD2014
7. Patients with Diabetes Type I or uncontrolled Type II (HbA1c >59 mmol/mol assessed locally) as judged by the investigator
8. Major surgery within 4 weeks prior to entry to the study (excluding placement of vascular access), or minor surgery within 2 weeks of entry into the study and from which the patient has not yet recovered
9. Treatment with warfarin. Patients on warfarin for DVT/PE can be converted to LMWH.
10. Potent and moderate inhibitors and inducers of CYP3A4/5 if taken within the stated washout periods:

    * Inhibitors (competitive): ketoconazole, itraconazole, indinavir, saquinovir, nelfinavir, atazanavir, amprenavir, fosamprenavir, troleandomycin, telithromycin, fluconazole, nefazodone, cimetidine, aprepitant, miconazole, fluvoxamine (1 week minimum wash-out period), amiodarone (27 week minimum wash-out period)
    * Inhibitors (time dependent): erythromycin, clarithromycin, verapamil, ritonavir, diltiazem (2 week minimum wash-out period)
    * Inducers: phenytoin, rifampicin, St. John's Wort, carbamazepine, primidone, griseofulvin, barbiturates, troglitazone, pioglitazone, oxcarbazepine, nevirapine, efavirenz, rifabutin (3 week minimum wash-out period) and phenobarbitone (5 week minimum washout period)
11. Potent and moderate inhibitors and inducers of CYP2C8 if taken within the stated washout periods:

    * Inhibitors: Gemfibrozil, trimethoprim, glitazones, montelukast, quercetin (1 week minimum wash-out period)
    * Inducers: Rifampicin (3 week minimum wash-out period)
12. At high medical risk because of non-malignant systemic disease including active uncontrolled infection e.g. interstitial lung disease, severe hepatic impairment, uncontrolled chronic renal disease
13. Known to be serologically positive for hepatitis B, hepatitis C or human immunodeficiency virus (HIV).
14. Patients who have experienced any of the following procedures or conditions currently or in the preceding 12 months:

    * coronary artery bypass graft
    * angioplasty
    * vascular stent
    * myocardial infarction (MI)
    * uncontrolled angina pectoris
    * congestive heart failure NYHA Grade 2
    * ventricular arrhythmias requiring continuous therapy
    * supraventricular arrhythmias including AF, which are uncontrolled
    * Torsades de Pointes
    * haemorrhagic or thrombotic stroke, including transient ischaemic attacks or any other central nervous system bleeding
15. Resting ECG with measurable QTc interval of >470ms msec at 2 or more time points within a 24 hour period.
16. Concomitant medications known to prolong QT interval, or with factors that increase the risk of QTc prolongation or risk of arrhythmic events (such as heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome), or unexplained sudden death under 40 years of age. Inability to discontinue medication with agents designated as having a risk of Torsades de Pointes due to QT prolongation (see Appendix 5)
17. Left ventricular (LV) dysfunction (LVEF outside institutional range of normal) by MUGA or Echocardiogram.
18. Current malignancies of other types, with the exception of adequately treated cone-biopsied in situ carcinoma of the cervix, uteri and basal or squamous cell carcinoma of the skin. Cancer survivors, who have undergone potentially curative therapy for a prior malignancy, have no evidence of that disease for three years or more and are deemed at negligible risk for recurrence, are eligible for the trial.
19. Prior bone marrow transplant or have had extensive radiotherapy to greater than 25% of bone marrow within eight weeks of starting trial
20. Patients participating in or planning to participate in another interventional clinical trial whilst on this study. Participation in an observational trial is acceptable.
21. Any other condition which in the Investigator's opinion would not make the patient a good candidate for the clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-04-26 (Actual); Primary Completion 2017-11-15 (Actual); Study Completion 2017-11-15 (Actual)

PRIMARY OUTCOMES:
Establish the maximum tolerated dose and recommended Phase II dose of two intermittent dosing schedules of AZD2014: 3 days on, 4 days off and 2 days on, 5 days off in combination with weekly paclitaxel in patients with solid tumours. | First cycle of treamtent (7 weeks)
  To determine the dose at which no more than one patient out of up to 6 patients at the same dose level experience a drug-related dose-limiting toxicity.

SECONDARY OUTCOMES:
PK parameters for AZD2014 and paclitaxel derived from determining their plasma concentrations using validated assays. | First cycle of treatment (7 weeks)
  To explore the effect of paclitaxel on the pharmacokinetics of AZD2014
PK parameters for AZD2014 and paclitaxel derived from determining their plasma concentrations using validated assays | First cycle of treatment (7 weeks)
  Investigate the pharmacodynamics behaviour of the combination of AZD2014 and paclitaxel.

OTHER OUTCOMES:
To document any possible anti-tumour activity | Duration of the study
  To determine disease response by RECIST criteria version 1.1, GCIG CA125 criteria and change in tumour size.

CONTACTS AND LOCATIONS:
Overall Officials: Udai Banerji, PhD, Principal Investigator — The Institute of Cancer Research, Royal Marsden NHS Foundation Trust
Locations (4):
- United Kingdom (4):
  - Addenbrookes Hospital, Cambridge, Cambridgeshire
  - Royal Marsden Hospital, Sutton, Surrey
  - Belfast City Hospital, Belfast
  - Guy's and St Thomas's NHS Foundation Trust, London

REFERENCES:
- [Background] Basu B, Krebs MG, Sundar R, Wilson RH, Spicer J, Jones R, Brada M, Talbot DC, Steele N, Ingles Garces AH, Brugger W, Harrington EA, Evans J, Hall E, Tovey H, de Oliveira FM, Carreira S, Swales K, Ruddle R, Raynaud FI, Purchase B, Dawes JC, Parmar M, Turner AJ, Tunariu N, Banerjee S, de Bono JS, Banerji U. Vistusertib (dual m-TORC1/2 inhibitor) in combination with paclitaxel in patients with high-grade serous ovarian and squamous non-small-cell lung cancer. Ann Oncol. 2018 Sep 1;29(9):1918-1925. doi: 10.1093/annonc/mdy245. PMID 30016392